CLINICAL TRIAL: NCT03148522
Title: Clinical Psychopharmacology Division,Institute of Mental Health,Peking University
Brief Title: A Diagnosis and Treatment Optimization Study of Depression Based on the Neurological Mechanism of Reward System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Si Tianmei, Director of Clinical Psychopharmacology Division Institute of Mental Health, Peking University, Peking University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 81630031
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Diagnosis and Treatment of Depression
MeSH Terms: conditions — Disease | interventions — Escitalopram; Duloxetine Hydrochloride; Mirtazapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- escitalopram (Experimental): Eligible patients were assigned to escitalopram treatment based on investigators' clinical practice.
  Interventions: Drug: Escitalopram
- duloxetine (Experimental): Eligible patients were assigned to duloxetine treatment based on investigators' clinical practice.
  Interventions: Drug: Duloxetine
- mirtazapine (Experimental): Eligible patients were assigned to mirtazapine treatment based on investigators' clinical practice.
  Interventions: Drug: Mirtazapine

INTERVENTIONS:
Drug: Escitalopram — receive escitalopram
  Arms: escitalopram
Drug: Duloxetine — receive duloxetine
  Arms: duloxetine
Drug: Mirtazapine — receive mirtazapine
  Arms: mirtazapine

SUMMARY:
Major depressive disorder (MDD) is a high-disabling disease. But its etiology and pathogenesis is not clear, and early recognition, diagnosis and treatment still has many challenges. Among numerous clinical manifestations of MDD, anhedonia is an important core symptom of MDD, especially in patients with melancholic features. Our previous studies and studies abroad have shown that MDD patients had functional abnormality in reward circuit. The abnormalities of reward-related core areas, such as the prefrontal cortex - nucleus accumbens - ventral tegmental area were closely associated with the development of MDD, and is an important neural basis of anhedonia. This study would take the reward circuit as mainline to carry out the etiology, diagnosis and therapeutic intervention studies of MDD. We would collect MDD patients with melancholic features and other populations with reward dysfunction. The neuroimaging techniques, stress assessment, genetic testing and drug intervention methods would be mainly used in this study. The functional connectivity of reward regions, such as the ventral striatum, nucleus accumben, and ventral medial prefrontal cortex, would be analyzed to identify the dysfunction of reward circuit of MDD, and its implication for early recognition, diagnosis and prediction of treatment efficacy of antidepressants. We would also investigate the effect of genetic and environmental factors on reward function of MDD and its biological basis. Finally, through modulating the reward circuit activity using animal experiments, we would verify and investigate reward dysfunction of MDD and its biological mechanisms. The project is expected to provide for new evidence for the establishment of reward mechanism - based objective diagnosis and treatment optimization strategy of MDD.

ELIGIBILITY:
Inclusion Criteria:

* first-episode, drug naive melancholic depression; remitted depression; schizophrenia patients; first-degree relatives of depressed patients.

Exclusion Criteria:

* major somatic diseases; DSM-IV axis I other mental illness; personality disorder, mental retardation; drug and / or alcohol dependence; serious suicidal tendencies or suicidal behavior; pregnant or lactating women; MRI contraindications.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression | 8 weeks
  remission defined by Hamilton Rating Scale for Depression < 7

CONTACTS AND LOCATIONS:
Locations (1):
- Yun-Ai SU, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin J, Su Y, Rizvi SJ, Jagoda J, Li J, Wu Y, Dai Y, Zhang Y, Kennedy SH, Si T. Define and characterize the anhedonia in major depressive disorder: An explorative study. J Affect Disord. 2022 Sep 15;313:235-242. doi: 10.1016/j.jad.2022.06.082. Epub 2022 Jul 3. PMID 35788366